CLINICAL TRIAL: NCT06129734
Title: Phase 1B/2A Study of Weekly Decitabine and Venetoclax Treatment as Maintenance Therapy in High-Risk Myeloid Malignancy Patients Post Allograft Stem Cell Transplant
Brief Title: Decitabine and Venetoclax Treatment as Maintenance Therapy in Patients Post Allograft Stem Cell Transplant
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Benjamin Tomlinson (Other)
Responsible Party: Sponsor-Investigator, Benjamin Tomlinson, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2923
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Myeloid Malignancy; Acute Myeloid Leukemia
Keywords: Allograft Stem Cell Transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low dose maintenance chemotherapy (Experimental): Participants will receive low dose chemotherapy as a maintenance therapy post-transplant. Participants must enroll by post-transplant day 40. Treatment will consist of once weekly 5 mg/m2 decitabine followed by 400 mg venetoclax orally approximately 6 hours afterwards. Participants will continue maintenance therapy for one year or unacceptable toxicity. Participants will otherwise receive post Allogeneic hematopoietic stem cell transplant (alloSCT) care and disease monitoring as per institutional standards.
  Interventions: Drug: Venetoclax; Drug: Decitabine

INTERVENTIONS:
Drug: Venetoclax — Venetoclax is a BCL2 inhibitor. It is administered at low doses and used in combination with other hypomethylating agents such as decitabine to manage participants with acute myeloid lymphoma who have undergone stem cell transplant. Participants will initiate therapy with decitabine that will be followed by venetoclax 400 mg oral 6-8 hours later. Participants will continue this dose each week. The venetoclax dose will be reduced to 100 mg once per week if the participant is being treated with posaconazole or voriconazole (strong CYP3A4 inhibitors) (considered dose equivalent to venetoclax 400 mg 1X/week). The venetoclax dose will be reduced 200 mg once per week if the participant is being treated with fluconazole or isavuconazole (moderate CYP3A4 inhibitors) (considered dose equivalent to venetoclax 400 mg 1X/week). This clinical trial is administering venetoclax well below the current FDA approved dosing.
Drug: Decitabine — Decitabine is a hypomethylating agent. It is administered at low doses and used in combination with venetoclax to manage participants with acute myeloid lymphoma who have undergone stem cell transplant. Participants initiate therapy with 5 mg/m2 decitabine subcutaneous every week followed by venetoclax.

SUMMARY:
The goal of this interventional clinical trial is to determine if low doses of gentle chemotherapy after bone marrow transplant may prevent relapse and promote an increase in survival and decrease in side effects in participants with acute myeloid leukemia and myelodysplastic syndromes. The main question it aims to answer is whether or not providing a new, gentler way of administering chemotherapy will help control leftover cancer with minimal side effects. This treatment involves decitabine and venetoclax. Participants will receive standard post-transplant care. Participants will be administered decitabine once per week with normal transplant follow up visits, and then will take a venetoclax pill about 6 to 8 hours later. Participants will meet their study team at the beginning, midway, and at the end of the trial to receive bone marrow testing. Participants will receive treatment until either one year of therapy, relapse, or recurrent dose limiting toxicity (DLT) despite dose reduction.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is the most common acute leukemia in adults. While 60-80% patients can achieve remission, a high rate of relapse mandates consolidative treatment. Unfortunately, 40% of AML patients and 30% of myelodysplastic syndrome patients will relapse after alloSCT, and those who relapse after transplant exhibit poor outcomes. As such, prevention of post-transplant relapse remains a key interest. Maintenance therapy with low-intensity chemotherapy and/or targeted therapy is one strategy that holds promise to reduce post-transplant relapse, controlling residual subclinical disease before frank relapse. As post-transplant maintenance strategies yield mixed results, standard of care maintenance therapy remains an unmet clinical need.

The combination of hypomethylating agents (HMAs), such as decitabine or 5-azacytidine, and the B-cell lymphoma 2 (BCL2) inhibitor venetoclax combination has transformed the management of transplant-ineligible AML patient improving median overall survival (OS) to 14.7 months compared to 9.6 months with azacytidine and placebo at the cost of more pronounced cytopenias (Grade 3 and 4 thrombocytopenia and neutropenia occurring in 45%/38% and 42%/28% respectively).

Recent work has demonstrated a mechanism by which HMAs cooperate with venetoclax, via priming AML cells for death via the integrated stress response (ISR). The ISR transcription factor activating transcription factor-4 (ATF4) is upregulated in a matter of hours after HMA treatment, and in turn activates Phorbol-12-myristate-13-acetate-induced protein 1 (PMAIP1) (NOXA) that degrades the BCL2-family member myeloid cell leukemia sequence 1 (MCL1), thus creating greater dependence in HMA-exposed malignant cells on BCL2 to avoid BAX/BAK mediated mitochondrial outer membrane permeabilization (MOMP), caspase release, and subsequent apoptosis. An irreversible step toward apoptosis is mitochondrial outer membrane permeabilization (MOMP) by BAX/BAK oligomers, which releases caspase proteases into the cells, a commitment into apoptosis that is fundamentally counteracted by BCL2-family antiapoptotic proteins, e.g., BCL2, the target of venetoclax inhibition. This mechanism primes AML blasts for venetoclax-mediated toxicity.

Through rigorous pharmacological optimization, it has been shown that the decitabine 5 mg/m2 weekly with a single dose of venetoclax 6 hours after the decitabine can control disease with limited effects normal hematopoietic cells.9 This novel dosing regimen may maximize decitabine/venetoclax anti-leukemic activity while minimizing hematologic toxicity and represents an attractive regimen for post-alloSCT maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute myeloid leukemia, MDS, MDS/AML with high-risk for post-transplant relapse identified by:

  * Very high or high risk by CIBMTR Disease Risk Index (DRI) and/or adverse risk by ICC 2022 criteria and/or MDS/AML by ICC 2022 criteria.
  * Very high or high risk by CIBMTR DRI and/or by IPSS-M > 0.510-12 and/or MDS/AML by ICC 2022 criteria.
* Bone marrow myeloblasts <5% at pre-transplant bone marrow aspirate and biopsy with no circulating blasts.
* Participants must be planned for or have received alloSCT. Any conditioning regimen intensity or graft source (MRD/MUD/Haplo/UCB) is permitted.
* Participants must be 18 years of age or older.
* Total bilirubin < 2.0 mg/dL (with the exception of participants with known Gilbert's syndrome, who should have direct bilirubin < 2 × ULN).
* Creatinine clearance (CrCl) > 30 ml/min.
* ECOG 0-1 performance status.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document and complete study related procedures.
* Participants may enroll prior to or after alloSCT. Participants should enroll no later than post transplant day 40, and the the following post-AlloHSCT inclusion criteria must be met in order to initiate the maintenance study treatment:

  * Successful engraftment defined by absolute neutrophil count (ANC) of ≥500/ul and platelet count of ≥50,000/uL sustained for at least three consecutive days.
  * These criteria for engraftment should be met on or before Day +50.
  * No active infection
  * No GVHD ≥ overall grade II (Grade 1 GVHD of the skin acceptable).
  * Participants must continue to meet additional inclusion criteria
  * <5% myeloblasts in a bone marrow aspirate with spicules, that is to be obtained, if all the above inclusion criteria are satisfied.

Exclusion Criteria:

* Prior disease progression on HMA/VEN therapy, single agent venetoclax.
* Other planned post-transplant maintenance therapy, such as FLT3-ITD targeting agents, as determined by the treating physician
* Currently pregnant or breast-feeding. Females of childbearing (FOCBP) potential must have negative serum pregnancy test within 72 hours from treatment start. (NOTE: FOCBP is any biologic female, regardless of sexual or gender orientation, having undergone tubal ligation, or remaining celibate by choice, who has not undergone a documented hysterectomy or bilateral oophorectomy or has had a menses any time in the preceding 12 months (therefore not naturally post-menopausal for > 12 months)
* Uncontrolled comorbid illness that could limit life expectancy or ability to complete study correlates. This includes, but is not limited to:

  * Active infection
  * Uncontrolled concurrent malignancy
  * Congestive heart failure of NYHA class III/IV. Participants with compensated heart failure are permitted.
  * Unstable angina pectoris
  * New or unstable cardiac arrhythmia. Stable or controlled arrhythmias are permitted
  * Decompensated liver cirrhosis (Child-Pugh score ≥12 or a MELD score ≥21
  * Psychiatric illness/social situations that would limit compliance with study requirements.
  * Any other prior or ongoing condition, in the opinion of the investigator, that could adversely affect the safety of the participants or impair the assessment of study results.
* FOCBP and males that are unwilling to agree to use dual contraceptive measures (i.e., hormonal or barrier method of birth control; abstinence, condom) prior to study entry and for the duration of study participation. Should a female subject become pregnant or suspect she is pregnant while participating in this study, they should inform the treating physician immediately
* Sexually active male who is unwilling to use a condom when engaging in any sexual contact with a female with child-bearing potential, beginning at the screening visit and continuing until 4 weeks after taking the last dose of decitabine/venetoclax.
* Participants with known active HIV infection, as this will further increase the risk for opportunistic infections. However, participants with chronic HIV with undetectable viral load by PCR, without opportunistic infection, and on a stable regimen of antiretroviral therapy would be eligible.
* Known allergy or hypersensitivity to any component of decitabine/venetoclax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by dose limiting toxicities | 1 year after treatment
  The primary objective of this study will be to assess the safety of low dose decitabine/venetoclax in the post transplant setting. Safety will be defined in accordance with FDA guidance on development for new therapeutics in AML with the particular criteria to be considered as DLTs.
  The stopping criteria are described for the incidence of dose limiting toxicities that are at least possibly related to the study treatment.
  Using Bayesian toxicity monitoring with maximum DLT probability as 0.15, prior distribution (0.5, 0.5), maximum participants 20, minimum number of participants before stopping 9, cohort size 5, and posterior probability 0.8, the study will be paused for review if (2, 3, 4, 5) or more participants experiencing such Grade 4 events in (69, 11, 16, 20) participants, respectively.
Feasibility as measured by the rate of participants receiving planned treatment | 1 year after treatment
  The primary objective of this study will be to assess the feasibility of low dose decitabine/venetoclax in the post transplant setting. Feasibility will be defined as ≥ 80% of participants receiving ≥80% of planned decitabine/venetoclax doses, excluding participants removed from the study in the event of relapse.

SECONDARY OUTCOMES:
Rate of relapse free survival | 1 year after treatment
  The secondary objective is to determine the effects of low dose decitabine/venetoclax on the one relapse free survival compared to CIBMTR historical Disease Risk Index (DRI) data. The CIBMTR Disease Risk Index (DRI) is a clinically validated tool to predict survival post-transplant survival.
  Relapse-free survival (RFS) is measured from the date of the stem cell infusion to the date of disease progression or the date of death, whichever occurs first; and is censored at the date of last followed for those alive without disease progression. Relapse will be defined as more than 5% blasts on bone marrow biopsy, or, in the case of myelodysplastic syndrome (MDS), any clinical change that in the treating physician's opinion triggers change in therapy and will be compared to historical CIBMTR controls for very high or high risk for relapse by CIBMTR Disease Risk Index (DRI).

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Tomlinson, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center; James Ignatz-Hoover, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center; Claudio Brunstein, MD, PhD, Principal Investigator — Cleveland Clinic Foundation, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Seidman Cancer, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant data that underlie or influence the results observed from the study
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Compiled and analyzed patient data will be published upon study completion. Publisher may request Protocol and Statistical Analysis Plan
Access Criteria: Investigators who provide a methodologically sound proposal for use of requested data